CLINICAL TRIAL: NCT05452499
Title: Pain Neuroscience Education and Therapeutic Exercise as a Treatment for Chronic Pain, Kinesiophobia and Increased Physical Functionality in Breast Cancer Survivors
Brief Title: Pain Neuroscience Education and Therapeutic Exercise as a Treatment for Breast Cancer Survivors Living With Sequelae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autónoma de Yucatán (Other)
Responsible Party: Principal Investigator, José Antonio Lores Peniche, Principal Investigator, Universidad Autónoma de Yucatán
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Folio No.03-2022
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Breast Neoplasms; Pain, Chronic; Kinesiophobia; Breast Cancer
Keywords: Breast neoplasms; Breast cancer survivors; Chronic pain; Pain; Kinesiophobia; Pain neuroscience education; Exercise
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain; Kinesiophobia; Pain; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Other: Pain neuroscience education and therapeutic exercise

INTERVENTIONS:
Other: Pain neuroscience education and therapeutic exercise — Participants will receive a 9-week physiotherapy program. Consisting of 3 sessions of pain neuroscience education and 24 sessions of therapeutic exercise (16 face-to-face sessions and 8 at home).

SUMMARY:
Introduction: Breast cancer represents the most common type of malignant neoplasm worldwide. Advances in diagnosis and treatment have increased the life expectancy of patients. However, the sequelae associated with treatment and disease in survivors such as chronic pain, kinesiophobia and loss of physical function represent a long-term health problem. Physical therapy is a frequently used strategy for the treatment of sequelae in the acute stage of the disease, but there is a need to evaluate its effectiveness in cancer survivors with chronic sequelae. Therapeutic exercise and pain neuroscience education have been shown to be effective in the management of populations with chronic pain and loss of function; however, more evidence is needed in specific populations of cancer survivors. Objective:To evaluate the effectiveness of a physical therapy program based on pain neuroscience education and therapeutic exercise for the treatment of chronic pain, kinesiophobia and loss of physical function in breast cancer survivors. Methodology. Quasi-experimental study. The sample will consist of 40 female breast cancer survivors. The intervention will last 9 weeks, with 3 sessions of pain neuroscience education and 24 sessions of therapeutic exercise, 3 times per week (16 face-to-face sessions and 8 sessions at home). The intervention will be carried out in small groups of 8 to 12 people. The frequency and intensity of pain, the level of kinesiophobia and physical functionality and the range of of motion of the shoulder will be evaluated in 4 assessments, before the intervention (T0), 3rd (T1), 6th (T2) and 9th (T3) week of the intervention. Different validated measurement instruments will be used in this population such as self-report scales, questionnaires and the use of a goniometer.

ELIGIBILITY:
Inclusion Criteria:

1. Have had a stage I to III diagnosis.
2. Report a pain intensity of 30 millimeters or more in the Visual Analoge Scale (VAS).
3. Be in completed remission and have completed primary treatment at least three months age. Adjuvant hormone therapy or inmunotherapy is accepted.
4. Present pain in the neck, arms or shoulder of the affected side after primary cancer treatment, and that is repeated or maintained for a period longer than three months.
5. Presenting kinesiophobia measured with the Tampa Scale for Kinesiophobia (TSK-11V).
6. That presents alterations in the physical functionality of the upper limb, measured with the Upper Limb Functional Index (ULFI-Sp).
7. Who is willing to participate through informed consent.

9. Due to the current health situation in a state of pandemic by COVID-19, the patient must have their full COVID-19 vaccination.

Exclusion Criteria:

1. That presents some other type of cancer or metastasis at the time of the study.
2. Have uncontrolled lymphedema or uncontrolled hypertension.
3. That presents a musculoskeletal pathology in the upper limb or a chronic health condition that limits the performance of the therapeutic exercise.
4. Difficulty understanding the Spanish language that limits the comprehension of the evaluation instruments or participating in the pain neuroscience education program.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Changes in pain intensity | Four evaluations will be performed, before the intervention (T0) and at the 3rd (T1), 6th (T2) and 9th (T3) week of the physiotherapy program.
  Pain intensity will be measured using the visual analog scale (VAS), participants will report their pain intensity within a range of 0 to 100 millimeters, with 0 being no pain and 100 being the maximum pain.
Changes in pain frequency | Four evaluations will be performed, before the intervention (T0) and at the 3rd (T1), 6th (T2) and 9th (T3) week of the physiotherapy program.
  Participants will report the number of days per week with pain.

SECONDARY OUTCOMES:
Changes in kinesiophobia | Four evaluations will be performed, before the intervention (T0) and at the 3rd (T1), 6th (T2) and 9th (T3) week of the physiotherapy program.
  Kinesiophobia will be measured through the Tampa Kinesiophobia Scale Spanish version with 11 items (TSK-11V). It consists of a self-report instrument with 11 items related to fear of movement or injury relapse. Each ítem is measured on a Likert-type scale between 1 and 4 points, being 1 totally disagree and 4 totally agree, being able to obtain a total between a range of 11 to 44 final points. The higher the score, the higher the level of kinesiophobia.
Changes in physical functionality | Four evaluations will be performed, before the intervention (T0) and at the 3rd (T1), 6th (T2) and 9th (T3) week of the physiotherapy program.
  Physical functionality will be measured through the Upper Limb Functional Index scale (ULFI-Sp), which consists of a list of 25 items. Each item is scored on a 3-point scale by filling in a box, so that filling in the whole box means strongly agree, half a box means partially agree, and leaving it empty means strongly disagree, giving it a score of 1, 0.5 and 0 points respectively. The total score (25 points maximum) is multiplied by 4 to obtain a score based on 100 points, of which 0 would represent no functional limitation and 100 maximum limitation. The first 16 items refer to common functional activities, while the other 9 focus on activities involving the use of the upper limb.
Shoulder range of motion | Four evaluations will be performed, before the intervention (T0) and at the 3rd (T1), 6th (T2) and 9th (T3) week of the physiotherapy program.
  Active joint range of motion (active ROM) will be measured as part of the physical function assessment of the patient's upper limb. Flexion, horizontal flexion, extension, internal rotation, external rotation and abduction of both shoulders will be measured. Active ROM will be measured using a BASELINE® brand 12-inch shoulder goniometer. Three goniometric measurements will be taken per movement, and the average will be taken to obtain a value of the active ROM between a range of 0 and 180 degrees.

OTHER OUTCOMES:
Personal characteristics | This data will be recollected only before the intervention (T0).
  An initial survey with 2 sections will be applied: the first will collect information on sociodemographic variables such as: age, marital status, occupation, level of schooling, weight, height, BMI, habits (alcohol and tobacco) and comorbidities. The second will contain questions on the clinical characteristics of breast cancer such as: number of months with pain, time since initial diagnosis, time elapsed and stage of breast cancer at diagnosis, type of breast cancer according to histological classification, hormone receptor status, location of breast cancer (right, left or bilateral), type of surgery and other treatments (radiotherapy, chemotherapy, hormone therapy or inmunotherapy), the region of pain (axilla, shoulder, arm or thorax).
Evaluation of neuropathic and nociceptive type of pain | Four evaluations will be performed, before the intervention (T0) and at the 3rd (T1), 6th (T2) and 9th (T3) week of the physiotherapy program.
  The DN4 questionnarie will be used to discriminate between neuropathic and nociceptive type of pain. The DN4 questionnaire consists of a total of 10 items grouped in 4 sections. The first seven items are related to the quality of pain (burning, painful cold, electric shocks) and its association to abnormal sensations (tingling, pins and needles, numbness, itching). The other 3 items are related to neurological examination in the painful area (touch hypoesthesia, pinprick hypoesthesia, tactile allodynia). A score of 1 is given to each positive item and a score of 0 to each negative item. The total score is calculated as the sum of all 10 items, and the cut-off value for the diagnosis of neuropathic pain is a total score of 4/10.
Central sensitization | Four evaluations will be performed, before the intervention (T0) and at the 3rd (T1), 6th (T2) and 9th (T3) week of the physiotherapy program.
  To evaluate central sensitization related symptoms part A of the Spanish Central Sensitization Inventory (CSI) will be used. Part A of the CSI assesses 25 health-related symptoms common to central sensitization, with total scores ranging from 0 to 100. . A total score of 40 or higher indicates the presence of central sensitization.
Evaluation of nociplastic type of pain. | Four evaluations will be performed, before the intervention (T0) and at the 3rd (T1), 6th (T2) and 9th (T3) week of the physiotherapy program.
  To evaluate possible nociplastic pain, the clinical criteria for nociplastic pain affecting the musculoeskeletal system propose by the International Association for The Study of Pain (IASP) Terminology Task Force (TTF) will be used. It consists of 4 items to clinically evaluate: the type of pain (if greater than 3 months, its distribution and the presence or not of nociceptive type of pain), history of hypersensitivity in the region of pain, presence of comorbidities (sensitivity to sound or light, sleep problems, fatigue or cognitive problems), evoked pain hypersensitivity in the region of pain (static mechanical allodynia, static dynamic allodynia, allodynia to heat or cold). Presence of item 1 and 4 is classifed as possible nociplastic pain, and all of the above (item 1, 2, 3 and 4) as probable nociplastic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Antonio Lores, PT, Principal Investigator — Universidad Autónoma de Yucatán
Locations (1):
- Jose Antonio Lores Peniche, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: Undecided